CLINICAL TRIAL: NCT02593539
Title: An Open-label, Single Arm Study to Investigate the Safety, Pharmacokinetics and Pharmacodynamics of Repeat Doses of Inhaled Nemiralisib in Patients With APDS/PASLI
Brief Title: Safety, Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of Repeat Doses of Inhaled Nemiralisib in Patients With APDS/PASLI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204745; 2015-004876-31 (EudraCT Number)
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Activated PI3K-delta Syndrome
Keywords: APDS; Safety; Pharmacokinetics; GSK2269557; PASLI
MeSH Terms: conditions — Activated PI3K-delta Syndrome | interventions — Nemiralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants recieving nemiralisib (Experimental)
  Interventions: Drug: Nemiralisib

INTERVENTIONS:
Drug: Nemiralisib — Participants will be administered nemiralisib

SUMMARY:
This is an open-label study conducted to investigate safety, pharmacokinetics and pharmacodynamics of repeat doses of inhaled nemiralisib (NEMI) in participants with activated phosphoinositide 3-kinase (PI3K) delta syndrome /p110 delta-activating mutation causing senescent T Cells, lymphadenopathy and immunodeficiency (APDS/PASLI)

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 or older at the time of signing the informed consent.
* Patients with a clinical phenotype consistent with APDS, including a history of recurrent (frequency greater than would be expected in an immunocompetent individual) ear, sinus or pulmonary infections, and who have a known type 1 APDS-associated genetic PI3K delta mutation (i.e. E1021K, N334K, E525K and C416R).
* Body weight >=45 kilograms (kg) and body mass index (BMI) >=18 kg/square meter (m^2) (inclusive)
* Male subject. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until completion of the follow-up telephone call at 1-2 weeks from last dose. Vasectomy with documentation of azoospermia. Male condom plus partner use of one of the following contraceptive options: 1. Contraceptive subdermal implant 2. Intrauterine device or intrauterine system 3. Combined estrogen and progestogen oral contraceptive, 4. Injectable progestogen 5. Contraceptive vaginal ring 6. Percutaneous contraceptive patches. This is an all inclusive list of those methods that meet the GSK definition of highly effective: having a failure rate of less than 1% per year when used consistently and, correctly and, when applicable, in accordance with the product label. For non-product methods (e.g. male sterility), the investigator determines what is consistent and correct use. The GlaxoSmithKline (GSK) definition is based on the definition provided by International Conference on Harmonisation (ICH).
* Female subject. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: 1. Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. 2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until completion of the follow-up telephone call at 1-2 weeks from last dose.
* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) >2xupper limit normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease except where hepatomegaly is identified by their clinician to be secondary to APDS, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Regular or chronic treatment with strong inhibitors of Cytochrome P450 (CYP) 3A4 and/or CYP2D6 (this includes some anti-epileptic treatments, macrolide antibiotics, oral antifungal treatments and anti-tuberculosis therapy are prohibited from the screening visit until the end of treatment visit. Where clinically appropriate, an alternative drug in the same class (or unrelated class) that is not a strong CYP3A4 and/or CYP2D6 inhibitor can, after signing informed consent, be substituted for the original strong inhibitor of these enzymes
* Use of unstable dosing regimen with intravenous (i.v.) immunoglobulin (Ig) /subcutaneous (s.c.) Ig in the last 6 months before screening. Stable maintenance immunoglobulin regimen, as per local practice, such as regular injections with a consistent dosing interval (e.g. monthly) is acceptable.
* Previous use of an mechanistic target of rapamycin (mTOR) antagonist (e.g. rapamycin, everolimus) or PI3K delta inhibitor (selective or non-selective PI3K inhibitors).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (~240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof (including lactose) or a history of drug or other allergy (including a milk protein allergy) that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* History of previous intolerance of the induced sputum procedure.
* Bronchoalveolar Lavage (BAL) sub study only: History of bronchospasm in response to the brochoscopy/BAL procedure
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dose of study medication in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* A positive test for human immunodeficiency virus (HIV) antibody.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label study conducted to investigate safety, pharmacokinetics and pharmacodynamics of repeat doses of inhaled nemiralisib (NEMI) in participants with activated phosphoinositide 3-kinase (PI3K) delta syndrome /p110 delta-activating mutation causing senescent T Cells, lymphadenopathy and immunodeficiency (APDS/PASLI)
Pre-assignment Details: Participants received either 1000 mcg NEMI DISKUS or 700 mcg NEMI ELLIPTA or 500 mcg NEMI ELLIPTA. All NEMI DISKUS and NEMI ELLIPTA dose levels were combined as All NEMI treatment group as there was no intent to compare two dose levels or devices. The study had protocol amendments to reflect changes in dose and device administration.
Groups:
- All NEMI: Participants were administered with either NEMI 1000 mcg using DISKUS DPI or NEMI 700 or 500 mcg using ELLIPTA DPI once daily in the morning. NEMI DISKUS and NEMI ELLIPTA were combined as All NEMI treatment group as there was no intent to compare two dose levels or devices.
Period: Overall Study
Arm/Group | All NEMI
Started | 5
Completed | 4
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-White/Caucasian/European Heritage | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) and Any Non-serious Adverse Events (Non-SAEs)
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician. Number of participants with any SAE and non-SAEs are presented.
Time Frame: Upto 7.5 months
Population: All Subjects Population consisted of all participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Participants
  Any non-SAE | 5
  Any SAE | 0

2. Primary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in participants in a semi-supine position after 5 minutes rest. Baseline value is defined as latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value. Not applicable (NA) indicates that standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56, 83 and 84
Population: All Subjects Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Millimeters of Mercury (mmHg)
  DBP, Day 14, n= 5 | 1.0 (6.44)
  DBP, Day 28, n= 4: number analyzed (Participants) | 4
  DBP, Day 28, n= 4 | 4.0 (6.98)
  DBP, Day 56, n= 4: number analyzed (Participants) | 4
  DBP, Day 56, n= 4 | 8.5 (5.80)
  DBP, Day 83, n= 4: number analyzed (Participants) | 4
  DBP, Day 83, n= 4 | 2.0 (4.40)
  DBP, Day 84 n= 1: number analyzed (Participants) | 1
  DBP, Day 84 n= 1 | 17.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.
  SBP, Day 14, n= 5 | -1.0 (3.67)
  SBP, Day 28, n= 4: number analyzed (Participants) | 4
  SBP, Day 28, n= 4 | 5.3 (8.54)
  SBP, Day 56, n= 4: number analyzed (Participants) | 4
  SBP, Day 56, n= 4 | 10.0 (9.31)
  SBP, Day 83, n= 4: number analyzed (Participants) | 4
  SBP, Day 83, n= 4 | 1.5 (3.51)
  SBP, Day 84, n= 1: number analyzed (Participants) | 1
  SBP, Day 84, n= 1 | 16.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.

3. Primary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in participants in a semi-supine position after 5 minutes rest. Baseline value is defined as latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value. NA indicates that standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56, 83 and 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Beats per minute
  Day 14, n= 5 | 3.2 (7.73)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 2.0 (10.86)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 6.8 (9.43)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 4.8 (7.76)
  Day 84 n= 1: number analyzed (Participants) | 1
  Day 84 n= 1 | 7.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.

4. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in participants in a semi-supine position after 5 minutes rest. . Baseline value is defined as latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value. NA indicates that standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56, 83 and 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Breaths per minute
  Day 14, n= 5 | 0.2 (2.28)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 0.8 (4.57)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 1.5 (5.26)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 1.0 (2.45)
  Day 84 n= 1: number analyzed (Participants) | 1
  Day 84 n= 1 | 2.0 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.

5. Primary Outcome: Change From Baseline in Body Temperature
Description: Temperature was measured in participants in a semi-supine position after 5 minutes rest. Baseline value is defined as latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value. NA indicates that standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56, 83 and 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Degrees celsius
  Day 14, n= 5 | 0.10 (0.158)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 0.17 (0.350)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 0.07 (0.171)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 0.17 (0.479)
  Day 84 n= 1: number analyzed (Participants) | 1
  Day 84 n= 1 | 0.50 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed.

6. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Mean Heart Rate
Description: Single 12-lead ECGs were recorded at indicated timepoints using an ECG machine that automatically calculated the heart rate. Baseline value is defined as latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Beats per minute
  Day 14, n= 5 | -1.0 (3.94)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | -0.8 (2.99)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 5.3 (7.54)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 1.0 (2.31)

7. Primary Outcome: Change From Baseline in PR Interval, QRS Duration, Uncorrected QT Interval, QT Corrected Interval-Fredericia Interval (QTcF) and QTc Corrected by Bazett's Formula (QTcB)
Description: Twelve lead ECGs were recorded at indicated timepoints. At each time point, ECG machine automatically measured QRS duration, uncorrected QT interval, QTcF interval and QTcB. Baseline value is defined as latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Milliseconds
  PR, Day 14, n= 5 | -2.2 (9.23)
  PR, Day 28, n= 4: number analyzed (Participants) | 4
  PR, Day 28, n= 4 | -4.8 (4.27)
  PR, Day 56, n= 4: number analyzed (Participants) | 4
  PR, Day 56, n= 4 | -3.3 (11.18)
  PR, Day 83, n= 4: number analyzed (Participants) | 4
  PR, Day 83, n= 4 | -6.0 (11.80)
  QRS Duration, Day 14, n= 5 | -5.6 (7.33)
  QRS Duration, Day 28, n= 4: number analyzed (Participants) | 4
  QRS Duration, Day 28, n= 4 | -4.5 (11.03)
  QRS Duration, Day 56, n= 4: number analyzed (Participants) | 4
  QRS Duration, Day 56, n= 4 | -6.5 (8.81)
  QRS Duration, Day 83, n= 4: number analyzed (Participants) | 4
  QRS Duration, Day 83, n= 4 | -6.0 (7.79)
  QT Interval, Day 14, n= 5 | -7.2 (10.66)
  QT Interval, Day 28, n= 4: number analyzed (Participants) | 4
  QT Interval, Day 28, n= 4 | -2.8 (28.89)
  QT Interval, Day 56, n= 4: number analyzed (Participants) | 4
  QT Interval, Day 56, n= 4 | -22.3 (16.01)
  QT Interval, Day 83, n= 4: number analyzed (Participants) | 4
  QT Interval, Day 83, n= 4 | -16.3 (9.74)
  QTcB, Day 14, n= 5 | -9.4 (4.93)
  QTcB, Day 28, n= 4: number analyzed (Participants) | 4
  QTcB, Day 28, n= 4 | -4.5 (22.55)
  QTcB, Day 56, n= 4: number analyzed (Participants) | 4
  QTcB, Day 56, n= 4 | -8.3 (24.55)
  QTcB, Day 83, n= 4: number analyzed (Participants) | 4
  QTcB, Day 83, n= 4 | -12.5 (8.19)
  QTcF, Day 14, n= 5 | -8.2 (4.32)
  QTcF, Day 28, n= 4: number analyzed (Participants) | 4
  QTcF, Day 28, n= 4 | -3.5 (24.09)
  QTcF, Day 56, n= 4: number analyzed (Participants) | 4
  QTcF, Day 56, n= 4 | -13.0 (19.92)
  QTcF, Day 83, n= 4: number analyzed (Participants) | 4
  QTcF, Day 83, n= 4 | -14.0 (7.79)

8. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected for the analysis of clinical parameters including ALT, ALP and AST. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | All NEMI
Number analyzed (Participants) | 5
International units per liter (IU/L)
  ALT, Day 14, n= 5 | 1.0 (2.12)
  ALT, Day 28, n= 4: number analyzed (Participants) | 4
  ALT, Day 28, n= 4 | 0.8 (1.71)
  ALT, Day 56, n= 4: number analyzed (Participants) | 4
  ALT, Day 56, n= 4 | 0.0 (1.63)
  ALT, Day 83, n= 4: number analyzed (Participants) | 4
  ALT, Day 83, n= 4 | 1.3 (7.50)
  AST, Day 14, n= 5 | -0.8 (1.48)
  AST, Day 28, n= 4: number analyzed (Participants) | 4
  AST, Day 28, n= 4 | 0.8 (2.22)
  AST, Day 56, n= 4: number analyzed (Participants) | 4
  AST, Day 56, n= 4 | -0.8 (4.79)
  AST, Day 83, n= 4: number analyzed (Participants) | 4
  AST, Day 83, n= 4 | -1.0 (7.70)
  ALP, Day 14, n= 5 | 2.6 (5.77)
  ALP, Day 28, n= 4: number analyzed (Participants) | 4
  ALP, Day 28, n= 4 | 3.8 (5.68)
  ALP, Day 56, n= 4: number analyzed (Participants) | 4
  ALP, Day 56, n= 4 | 7.5 (5.00)
  ALP, Day 83, n= 4: number analyzed (Participants) | 4
  ALP, Day 83, n= 4 | 6.0 (2.94)

9. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters : Albumin and Total Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameter-albumin and total protein. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Grams per liter
  Albumin, Day 14, n= 5 | 2.6 (2.07)
  Albumin, Day 28, n= 4: number analyzed (Participants) | 4
  Albumin, Day 28, n= 4 | 1.3 (3.20)
  Albumin, Day 56, n= 4: number analyzed (Participants) | 4
  Albumin, Day 56, n= 4 | 2.8 (2.36)
  Albumin, Day 83, n= 4: number analyzed (Participants) | 4
  Albumin, Day 83, n= 4 | 2.0 (3.16)
  Total Protein, Day 14, n= 5 | 4.0 (1.58)
  Total Protein, Day 28, n= 4: number analyzed (Participants) | 4
  Total Protein, Day 28, n= 4 | 1.3 (3.59)
  Total Protein, Day 56, n= 4: number analyzed (Participants) | 4
  Total Protein, Day 56, n= 4 | 4.0 (4.76)
  Total Protein, Day 83, n= 4: number analyzed (Participants) | 4
  Total Protein, Day 83, n= 4 | 4.3 (2.50)

10. Primary Outcome: Change From Baseline Values in Clinical Chemistry Parameters: Sodium, Potassium, Calcium, Glucose and Urea
Description: Blood samples were collected for the analysis of clinical parameters including sodium, potassium, calcium, glucose and urea. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Millimoles per liter
  Sodium, Day 14, n= 5 | -0.2 (2.68)
  Sodium, Day 28, n= 4: number analyzed (Participants) | 4
  Sodium, Day 28, n= 4 | 0.5 (0.58)
  Sodium, Day 56, n= 4: number analyzed (Participants) | 4
  Sodium, Day 56, n= 4 | -0.8 (2.06)
  Sodium, Day 83, n= 4: number analyzed (Participants) | 4
  Sodium, Day 83, n= 4 | 0.0 (1.83)
  Potassium, Day 14, n= 5 | 0.24 (0.397)
  Potassium, Day 28, n= 4: number analyzed (Participants) | 4
  Potassium, Day 28, n= 4 | 0.30 (0.346)
  Potassium, Day 56, n= 4: number analyzed (Participants) | 4
  Potassium, Day 56, n= 4 | 0.35 (0.370)
  Potassium, Day 83, n= 4: number analyzed (Participants) | 4
  Potassium, Day 83, n= 4 | 0.38 (0.275)
  Calcium, Day 14, n= 5 | 0.040 (0.0990)
  Calcium, Day 28, n= 4: number analyzed (Participants) | 4
  Calcium, Day 28, n= 4 | 0.063 (0.0704)
  Calcium, Day 56, n= 4: number analyzed (Participants) | 4
  Calcium, Day 56, n= 4 | 0.133 (0.1343)
  Calcium, Day 83, n= 4: number analyzed (Participants) | 4
  Calcium, Day 83, n= 4 | 0.082 (0.1325)
  Glucose, Day 14, n= 5 | -0.64 (1.557)
  Glucose, Day 28, n= 4: number analyzed (Participants) | 4
  Glucose, Day 28, n= 4 | -0.60 (1.774)
  Glucose, Day 56, n= 4: number analyzed (Participants) | 4
  Glucose, Day 56, n= 4 | -0.48 (1.578)
  Glucose, Day 83, n= 4: number analyzed (Participants) | 4
  Glucose, Day 83, n= 4 | -0.68 (1.333)
  Urea, Day 14, n= 5 | 4.732 (5.8283)
  Urea, Day 28, n= 4: number analyzed (Participants) | 4
  Urea, Day 28, n= 4 | 8.330 (2.6837)
  Urea, Day 56, n= 4: number analyzed (Participants) | 4
  Urea, Day 56, n= 4 | 2.610 (5.1954)
  Urea, Day 83, n= 4: number analyzed (Participants) | 4
  Urea, Day 83, n= 4 | 2.185 (4.1025)

11. Primary Outcome: Change From Baseline Values in Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters: direct bilirubin, total bilirubin and creatinine. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Micromoles per liter
  Direct bilirubin, Day 14, n= 5 | -1.0 (0.71)
  Direct bilirubin, Day 28, n= 4: number analyzed (Participants) | 4
  Direct bilirubin, Day 28, n= 4 | -1.8 (0.96)
  Direct bilirubin, Day 56, n= 4: number analyzed (Participants) | 4
  Direct bilirubin, Day 56, n= 4 | -0.5 (1.00)
  Direct bilirubin, Day 83, n= 4: number analyzed (Participants) | 4
  Direct bilirubin, Day 83, n= 4 | -0.5 (1.00)
  Total bilirubin, Day 14, n= 5 | -1.8 (1.64)
  Total bilirubin, Day 28, n= 4: number analyzed (Participants) | 4
  Total bilirubin, Day 28, n= 4 | -3.0 (2.45)
  Total bilirubin, Day 56, n= 4: number analyzed (Participants) | 4
  Total bilirubin, Day 56, n= 4 | -0.8 (1.89)
  Total bilirubin, Day 83, n= 4: number analyzed (Participants) | 4
  Total bilirubin, Day 83, n= 4 | -1.5 (2.52)
  Creatinine , Day 14, n= 5 | -2.0 (12.43)
  Creatinine , Day 28, n= 4: number analyzed (Participants) | 4
  Creatinine , Day 28, n= 4 | -4.3 (6.08)
  Creatinine , Day 56, n= 4: number analyzed (Participants) | 4
  Creatinine , Day 56, n= 4 | 5.0 (14.07)
  Creatinine , Day 83, n= 4: number analyzed (Participants) | 4
  Creatinine , Day 83, n= 4 | -2.5 (14.93)

12. Primary Outcome: Change From Baseline Values in Clinical Chemistry Parameter: C-Reactive Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameter:C-Reactive Protein. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Milligrams per liter
  Day 14, n= 5 | 0.56 (1.592)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 0.75 (1.085)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 2.75 (6.222)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 3.90 (7.141)

13. Primary Outcome: Change From Baseline for Hematology Parameters: Basophil, Eosinophils, White Blood Cells (WBC), Lymphocytes, Neutrophils, Monocytes and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, WBC, lymphocytes, neutrophils, monocytes and platelets at indicated timepoints. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells per liters
Arm/Group | All NEMI
Number analyzed (Participants) | 5
10^9 cells per liters
  Basophils, Day 14, n= 5 | -0.002 (0.0045)
  Basophils, Day 28, n= 4: number analyzed (Participants) | 4
  Basophils, Day 28, n= 4 | 0.008 (0.0096)
  Basophils, Day 56, n= 4: number analyzed (Participants) | 4
  Basophils, Day 56, n= 4 | 0.008 (0.0236)
  Basophils, Day 83, n= 4: number analyzed (Participants) | 4
  Basophils, Day 83, n= 4 | 0.013 (0.0222)
  Eosinophils, Day 14, n= 5 | 0.108 (0.1542)
  Eosinophils, Day 28, n= 4: number analyzed (Participants) | 4
  Eosinophils, Day 28, n= 4 | 0.088 (0.0650)
  Eosinophils, Day 56, n= 4: number analyzed (Participants) | 4
  Eosinophils, Day 56, n= 4 | 0.128 (0.2241)
  Eosinophils, Day 83, n= 4: number analyzed (Participants) | 4
  Eosinophils, Day 83, n= 4 | 0.075 (0.0810)
  Lymphocytes, Day 14, n= 5 | 0.122 (0.2411)
  Lymphocytes, Day 28, n= 4: number analyzed (Participants) | 4
  Lymphocytes, Day 28, n= 4 | -0.133 (0.0918)
  Lymphocytes, Day 56, n= 4: number analyzed (Participants) | 4
  Lymphocytes, Day 56, n= 4 | -0.105 (0.1115)
  Lymphocytes, Day 83, n= 4: number analyzed (Participants) | 4
  Lymphocytes, Day 83, n= 4 | 0.037 (0.3140)
  Monocytes, Day 14, n= 5 | 0.096 (0.2893)
  Monocytes, Day 28, n= 4: number analyzed (Participants) | 4
  Monocytes, Day 28, n= 4 | 0.030 (0.0572)
  Monocytes, Day 56, n= 4: number analyzed (Participants) | 4
  Monocytes, Day 56, n= 4 | 0.115 (0.0614)
  Monocytes, Day 83, n= 4: number analyzed (Participants) | 4
  Monocytes, Day 83, n= 4 | 0.065 (0.0592)
  Neutrophils , Day 14, n= 5 | 0.334 (1.2388)
  Neutrophils , Day 28, n= 4: number analyzed (Participants) | 4
  Neutrophils , Day 28, n= 4 | 0.575 (0.6125)
  Neutrophils , Day 56, n= 4: number analyzed (Participants) | 4
  Neutrophils , Day 56, n= 4 | 0.553 (0.7647)
  Neutrophils , Day 83, n= 4: number analyzed (Participants) | 4
  Neutrophils , Day 83, n= 4 | 0.653 (0.7857)
  Platelet, Day 14, n= 5 | 49.4 (52.53)
  Platelet, Day 28, n= 4: number analyzed (Participants) | 4
  Platelet, Day 28, n= 4 | 9.0 (25.86)
  Platelet, Day 56, n= 4: number analyzed (Participants) | 4
  Platelet, Day 56, n= 4 | 17.0 (31.79)
  Platelet, Day 83, n= 4: number analyzed (Participants) | 4
  Platelet, Day 83, n= 4 | 61.8 (43.41)
  WBC, Day 14, n= 5 | 0.656 (1.0304)
  WBC, Day 28, n= 4: number analyzed (Participants) | 4
  WBC, Day 28, n= 4 | 0.568 (0.6004)
  WBC, Day 56, n= 4: number analyzed (Participants) | 4
  WBC, Day 56, n= 4 | 0.698 (1.0605)
  WBC, Day 83, n= 4: number analyzed (Participants) | 4
  WBC, Day 83, n= 4 | 0.845 (0.6608)

14. Primary Outcome: Change From Baseline for Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter: hemoglobin at indicated timepoints. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Grams per liter
  Day 14, n= 5 | 10.0 (5.24)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 8.3 (3.77)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 13.5 (8.50)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 13.3 (5.74)

15. Primary Outcome: Change From Baseline for Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit at indicated timepoints. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Percentage of red blood cells in blood
  Day 14, n= 5 | 0.0320 (0.01488)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 0.0333 (0.01204)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 0.0518 (0.02337)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 0.0465 (0.01396)

16. Primary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of hematology parameter: MCV at indicated timepoints. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Femtoliters
  Day 14, n= 5 | 1.00 (2.187)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 2.33 (2.287)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 2.02 (2.331)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 1.03 (3.407)

17. Primary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for the analysis of hematology parameters including MCH at indicated timepoints. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Picograms
  Day 14, n= 5 | 0.10 (0.485)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | -0.15 (0.676)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | -0.43 (0.763)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | -0.47 (0.525)

18. Primary Outcome: Change From Baseline for Hematology Parameter: Red Blood Cell Count
Description: Blood samples were collected for the analysis of hematology parameter: Blood Cell Count at indicated timepoints. Baseline value is defined as latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and at Days 14, 28, 56 and 83
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | All NEMI
Number analyzed (Participants) | 5
10^12 cells per liter
  Day 14, n= 5 | 0.304 (0.1417)
  Day 28, n= 4: number analyzed (Participants) | 4
  Day 28, n= 4 | 0.280 (0.0673)
  Day 56, n= 4: number analyzed (Participants) | 4
  Day 56, n= 4 | 0.488 (0.1640)
  Day 83, n= 4: number analyzed (Participants) | 4
  Day 83, n= 4 | 0.485 (0.1034)

19. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is used to assess pulmonary function using a spirometer at indicated timepoints. Baseline value is defined as the maximum measurement of the planned pre-dose measurements on Day 1, predose. Change from Baseline is defined as post-dose visit value minus Baseline value. Spirometry assessments were performed in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines
Time Frame: Baseline (Day 1: pre-dose) and at Day 1: 1 Hour post-dose; Day 2: 1 Hour post-dose; Day 14: Pre-dose; Day 14: 1 Hour post-dose and Day 83: Pre-dose
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | All NEMI
Number analyzed (Participants) | 5
Liters
  Day 1, 1 Hour post-dose: number analyzed (Participants) | 4
  Day 1, 1 Hour post-dose | 0.226 (0.2166)
  Day 2, 1 Hour post-dose: number analyzed (Participants) | 4
  Day 2, 1 Hour post-dose | 0.290 (0.2884)
  Day 14, Pre-dose: number analyzed (Participants) | 4
  Day 14, Pre-dose | -0.165 (0.5024)
  Day 14, 1 Hour post-dose | 0.016 (0.4812)
  Day 83, Pre-dose | -0.002 (0.4584)

20. Secondary Outcome: Plasma Concentration Following Administration of NEMI
Description: Blood samples for pharmacokinetic analysis was collected at the indicated time points following administration of NEMI. NA indicates that standard deviation could not be calculated as a single participant was analyzed
Time Frame: Day 1: Pre-dose, 5 minutes, 3 hours and 24 hours post-dose; Days 14 and 83: pre-dose
Population: Pharmacokinetic (PK) Population consisted of all participants in the 'All Subjects' population who had at least 1 non-missing PK assessment. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Groups:
- NEMI 1000 mcg Via DISKUS: Participants were administered NEMI 1000 mcg using DISKUS DPI once daily in the morning.
- NEMI 700 mcg Via ELLIPTA: Participants were administered NEMI 700 mcg using ELLIPTA DPI once daily in the morning.
- NEMI 500 mcg Via ELLIPTA: Participants were administered NEMI 500 mcg using ELLIPTA DPI once daily in the morning.
Arm/Group | NEMI 1000 mcg Via DISKUS | NEMI 700 mcg Via ELLIPTA | NEMI 500 mcg Via ELLIPTA
Number analyzed (Participants) | 1 | 1 | 3
Picograms per milliliter
  Day 1: Pre-dose; n=1,1,3 | 0.00 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 0.00 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 0.00 (0.00)
  Day 1: 5 minutes post-dose; n=1,1,3 | 467.00 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 1524.70 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 658.27 (394.468)
  Day 1: 3 hours post-dose; n=1,1,3 | 895.10 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 568.60 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 397.07 (172.226)
  Day 1: 24 hours post-dose; n=1,1,3 | 444.40 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 304.90 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 198.17 (82.442)
  Day 14: Pre-dose; n=1,1,3 | 1396.70 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 1242.60 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 750.83 (526.337)
  Day 83: Pre-dose; n=0,1,3: number analyzed (Participants) | 0 | 1 | 3
  Day 83: Pre-dose; n=0,1,3 |  | 1419.60 (NA) — NA indicates that standard deviation could not be calculated as a single participant was analyzed | 1525.83 (1181.340)

ADVERSE EVENTS:
Time Frame: Non-serious and serious adverse events were collected up to 7.5 months
Description: Non-serious and serious adverse events were collected in the All Subjects population. NEMI DISKUS and NEMI ELLIPTA were combined as All NEMI treatment group as there was no intent to compare two dose levels or devices.
Arm/Group | All NEMI
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All NEMI (N=5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Chest discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Feeling of body temperature change (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (7)
Oral candidiasis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 3 (22)
Migraine (Nervous system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Product taste abnormal (Product Issues) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT02593539/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT02593539/SAP_001.pdf